CLINICAL TRIAL: NCT05851755
Title: Italian Lung Cancer Observational Study
Acronym: LUCENT
Status: Enrolling by invitation | Type: Observational
Sponsor: The Mediterranean Institute for Transplantation and Advanced Specialized Therapies (Other)
Collaborators: S. Andrea Hospital (Other); Azienda Policlinico Umberto I (Other); Azienda Ospedaliero, Universitaria Pisana (Other); Università degli Studi dell'Aquila (Other); University of Milan (Other); Azienda Ospedaliera di Perugia (Other); Monaldi Hospital (Other); Azienda Ospedaliera di Bolzano (Other); AUSL Romagna Rimini (Other); European Institute of Oncology (Other); Università degli Studi di Ferrara (Other); Azienda Socio Sanitaria Territoriale di Mantova (Other)
Responsible Party: Sponsor
Other Study IDs: IRRB/04/23
Record Dates: First submitted 2023-04-30; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-04

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
LUCENT is an observational study focused on malignant pulmonary and tracheo-bronchial disease. It involves a large proportion of reference Italian thoracic surgery centers. The relevance of the study is related to the epidemiology of lung cancer in the world - also known as "Big Killer" - and the high mortality rates both in males and females.

The aim of his prospective study is to collect a large bulk of postoperative patients' outcome data and to produce up-to-date descriptive statistics of patients undergoing surgery for lung cancer. These results will be pivotal to compare the clinical results of all the relevant specialities involved in the care of lung cancer such as medical oncologists and radiation oncologists.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lung cancer
* informed consent

Exclusion Criteria:

* alcohol or drug abuse
* age < 18
* inability to express consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PaTientsin with lung cancer and an indication for respective surgery
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Lung cancer surgery outcomes | 5 years
  Benchmarking national outcome data of the treatment of lung cancer

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Crisci, MD, Principal Investigator — University of Aquila; Luca Bertolaccini, MD, Principal Investigator — European Institute of Oncology; Alessandro Bertani, MD, Principal Investigator — IRCCS ISMETT -UPMC ITALY
Locations (1):
- University of L'Aquila, L’Aquila, Italy

REFERENCES:
- [Derived] Bertolaccini L, Ciani O, Lucchi M, Zaraca F, Bertani A, Crisci R, Spaggiari L; LUCENT Study Group. Outcomes of Patients With Early and Locally Advanced Lung Cancer: Protocol for the Italian Lung Cancer Observational Study (LUCENT). JMIR Res Protoc. 2024 Oct 8;13:e57183. doi: 10.2196/57183. PMID 39378423